CLINICAL TRIAL: NCT05470231
Title: Effects of Beetroot Juice Intake on Repeated Performance of Elite Swimmers. A Randomized Controlled Study
Brief Title: Effect of Beet Juice on Elite Swimmers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Berta Moreno Heredero, PhD Sudent, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 42/2021
Record Dates: First submitted 2022-07-05; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: ergogéniques
Keywords: Swimming; Beetroot juice; Performance; Ergogenic aid

STUDY DESIGN:
Intervention Model Description: Parallel allocation was carried out in the two groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple blinded (Participant, Investigator and Outcomes Assessor) The participant was blinded not knowing the treatment to which he was submitted, investigator and outcome assessor responsible for collecting the results, without commenting on the group from which the subject came.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Active Comparator): The swimmers ingested a shot of Beet-It 70 ml beetroot juice (BJ)) 3 hours before undergoing a 6x100m crawl intermittent maximal speed performance test.
  Interventions: Dietary Supplement: Beetroot Juice
- Placebo (Placebo Comparator): The swimmers ingested a shot of Beet-It (70 ml placebo (PL)) 3 hours before undergoing a 6x100m crawl intermittent maximal speed performance test.
  Interventions: Dietary Supplement: Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — The swimmers drank 3 hours before the test, mL70 of BJ (containing mmol6.4 of NO-3) (Beet-It-Pro Elite Shot, James White Drinks Ltd., Ipswich, UK) or PLA (0.04 mmol of NO-3)

SUMMARY:
Objective: To investigate whether an acute intake of Beetroot Juice (BJ) improved performance factors in a repeated swimming effort at maximum speed in elite swimmers.

Methods: A total of 13 elite swimmers (6 girls and 7 boys) participated in this randomised, double-blind study. In 2 different trials, the swimmers ingested an injection of Beet-It (70 ml placebo (PL) or an injection of Beet-It 70 ml beetroot juice (BJ)) 3 hours before undergoing a 6x100m crawl intermittent maximal speed performance test.

ELIGIBILITY:
Inclusion Criteria:

* national and international level swimmers
* healthy swimmers
* no breakfast
* 48 hours with restricted diet of: other sports supplements and beetroot-rich foods

Exclusion Criteria:

* be on medication
* having had breakfast
* have brushed your teeth

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-01-25 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Lactate concentration | 3 hours post-dose of Beetroot juice or Placebo
  After the swimmers exited the water, their finger was wiped dry and their blood lactate concentration was measured with a portable Lactate Pro2 analyzer 1 minute after completing each 100-meter set.
Rate of Perceived Exertion | 3 hours after ingestion of the beetroot juice
  During the break between 100 and 100, they were asked how hard the effort had been using the subjective RPE scale as in other studies with BJ and swimming.
Recovery Total Quality Scale | 3 hours after ingestion of the beetroot juice
  Just before these same swimmers performed the next 100, they were asked how recovered they felt, using another subjective TQR scale
Total Time | 3 hours after ingestion of the beetroot juice
  The complete 6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the total times, with the program KINOVEA 0.9.5.
Parcial Time | 3 hours after ingestion of the beetroot juice
  The complete 6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the split times, with the KINOVEA 0.9.5 program.
Counter Movement Jump | 3 hours after ingestion of the beetroot juice
  Swimmers completed three repetitions of CMJ with hands on waist using an infrared jumping system (Optojump Next, Microgate, Bolzano, Italy)

SECONDARY OUTCOMES:
Stroke rate | from the day of randomization to the last day of the intervention: up to day 18
  The complete 6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the stroke rate, with the KINOVEA 0.9.5 program.
Underwater distance | from the day of randomization to the last day of the intervention: up to day 18
  The complete 6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the distances of the underwater swim at the start and the second turn, with the program KINOVEA 0.9.5.
Underwater time | from the day of randomization to the last day of the intervention: up to day 18
  The complete 6x100 main test was recorded with a JVC model GY-HM150E video camera placed on the stand of the facility itself at about 10 m from the start/turn wall (approximately 5 m above and 10 m from the swim lane) to record the entire session. The recording of the session made it possible to calculate the underwater time, with the KINOVEA 0.9.5 program.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Pozuelo de Alarcón, Spain

REFERENCES:
- [Background] Maughan RJ, Burke LM, Dvorak J, Larson-Meyer DE, Peeling P, Phillips SM, Rawson ES, Walsh NP, Garthe I, Geyer H, Meeusen R, van Loon LJC, Shirreffs SM, Spriet LL, Stuart M, Vernec A, Currell K, Ali VM, Budgett RG, Ljungqvist A, Mountjoy M, Pitsiladis YP, Soligard T, Erdener U, Engebretsen L. IOC consensus statement: dietary supplements and the high-performance athlete. Br J Sports Med. 2018 Apr;52(7):439-455. doi: 10.1136/bjsports-2018-099027. Epub 2018 Mar 14. PMID 29540367
- [Background] Dominguez R, Mate-Munoz JL, Cuenca E, Garcia-Fernandez P, Mata-Ordonez F, Lozano-Estevan MC, Veiga-Herreros P, da Silva SF, Garnacho-Castano MV. Effects of beetroot juice supplementation on intermittent high-intensity exercise efforts. J Int Soc Sports Nutr. 2018 Jan 5;15:2. doi: 10.1186/s12970-017-0204-9. eCollection 2018. PMID 29311764
- [Background] Lopez-Samanes A, Perez-Lopez A, Moreno-Perez V, Nakamura FY, Acebes-Sanchez J, Quintana-Milla I, Sanchez-Oliver AJ, Moreno-Perez D, Fernandez-Elias VE, Dominguez R. Effects of Beetroot Juice Ingestion on Physical Performance in Highly Competitive Tennis Players. Nutrients. 2020 Feb 23;12(2):584. doi: 10.3390/nu12020584. PMID 32102263
- [Background] Veiga S, Pla R, Qiu X, Boudet D, Guimard A. Effects of Extended Underwater Sections on the Physiological and Biomechanical Parameters of Competitive Swimmers. Front Physiol. 2022 Jan 26;13:815766. doi: 10.3389/fphys.2022.815766. eCollection 2022. PMID 35177993
- [Background] Tan R, Cano L, Lago-Rodriguez A, Dominguez R. The Effects of Dietary Nitrate Supplementation on Explosive Exercise Performance: A Systematic Review. Int J Environ Res Public Health. 2022 Jan 11;19(2):762. doi: 10.3390/ijerph19020762. PMID 35055584
- [Background] Senefeld JW, Wiggins CC, Regimbal RJ, Dominelli PB, Baker SE, Joyner MJ. Ergogenic Effect of Nitrate Supplementation: A Systematic Review and Meta-analysis. Med Sci Sports Exerc. 2020 Oct;52(10):2250-2261. doi: 10.1249/MSS.0000000000002363. PMID 32936597